CLINICAL TRIAL: NCT05640505
Title: Effectiveness of Gratitude Interventions for Academic Stress and Emotional Experiences Among Pakistani Adolescents
Brief Title: Gratitude Interventions for Academic Stress Among Pakistani Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Najam us Sahar, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UM.TNC2/UMREC-621
Record Dates: First submitted 2022-08-26; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Stress, Psychological
Keywords: Academic Expectations; Emotional Experiences
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Experimental research design with randomized control trial with difference of 4 weeks were be applied. Pretest post-test was done to compare the difference in the scores of academic stress and emotional experiences among adolescents before and after the intervention. Two experimental conditions will be used: (1) Gratitude (individuals assigned with daily gratitude-inducing activity) and (2) Control (no-assigned activity). Both groups were measured at (a) Pre-test (prior to the intervention); (b) Post-test (immediately after intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): This group received 03 gratitude interventions for 4 weeks
  Interventions: Behavioral: School based Gratitude Interventions
- Control Group (No Intervention): This group did not receive any intervention during active phase. Only the scores on dependent variables were measured. After completion of study, the same interventions were repeated with this group.

INTERVENTIONS:
Behavioral: School based Gratitude Interventions — Three gratitude interventions including Count your blessings, Gratitude Letter and Loving Kindness Meditation were applied with modification focusing on school related experiences. For example, writing a gratitude letter to a teacher, mentor or coach who played a significant role in one's life then imagining on the same person during LKM exercise of imagery. There were 9 sessions with 3-4 exercises in each session.
  Arms: Experimental

SUMMARY:
The experimental nature of this study will provide the empirical data in analyzing the effectiveness of gratitude exercises which later can be adapted in stress reduction programs at school level. This research will focus on the school related positive life experiences for example thinking about a teacher/mentor kindness and contribution in their lives, then write a letter that describes their gratitude & letter will be delivered to that person indirectly. This may help in focusing on the positive aspects of school life. This modification will serve as testing this new model for assessing the combined effect of gratitude interventions.

DETAILED DESCRIPTION:
Academic stress is an inevitable part of students' lives with long-term negative consequences on physical health, mental well-being, and social relations. In Asian cultures, expectations of parents and teachers are additional components of academic stress which have not been addressed in different stress management programs. Therefore, the present research addresses these contributory stress factors by using gratitude interventions in Pakistani high schools.

The study employs Broaden and Build Theory and Cognitive Appraisal Theory in formulating the intervention model and variables being tested through pretest-posttest experimental research design with a control group. A total of 102 high school students from two genders segregated schools of Rawalpindi city, Pakistan, served as the participants. They were randomly assigned into experimental and control groups, with 51 participants in each group. There were 41 boys and 61 girls with a mean age of 15.71+ 0.92 years. The measures included Academic Expectations Stress Inventory (AESI), Inventory of High-School Students' Recent Life Experiences (IHSSRLE), Modified Differential Emotions Scale (mDES), Gratitude Questionnaire-6 (GQ-6) and Gratitude Adjective Checklist (GAC). Three gratitude interventions, including Count your Blessings, Gratitude Letters and Loving-Kindness Meditation, were modified to focus on school-related experiences. The model consisted of nine sessions applied in schools for four weeks with 30-40 minutes each day. The research protocol and intervention model were adapted into Urdu for better understanding among participants. The data were analyzed through descriptive and inferential statistics (frequency, percentage, mean, SD, paired sample t-test, independent sample t-test, multivariate analysis of variance and effect size).

ELIGIBILITY:
Inclusion Criteria:

* High School Students
* Studying in same school for at least last six months
* within 14-17 years of age
* not having severe physical health issue or going under treatment for chronic illness

Exclusion Criteria:

* not able to understand Urdu language
* above 17 years of age or below 14 years
* recently enrolled in the particular school

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Academic Stress | 4 weeks
  Academic Expectations, Daily Hassles. Academic Expectation Stress Inventory is a nine (09) item inventory developed by Ang and Huan (Ang, Huan 2006) is a reliable and valid instrument widely used especially in assessing parental expectations (Ang et al., 2009; Qadir et al., 2012; Sun, 2012; Zhang et al., 2016). The two subscales are Self-Expectations and Other expectations covering the domains of stress, self-blame, disappointment, anxiety, and feeling of inadequacy. It has Likert - type scoring ranging from 1 (never true) to 5 (almost always true) with high scores showing more stress.
Emotional Experiences | 4 weeks
  Positive Emotions, Positivity Ratio. it will be measured through Modified Differential Emotions Scale is a reliable & valid instrument to assess positive and negative emotions separately.It is a twenty (20) items instrument with Five (05) points likert scoring from "Not at all" to "Extremely". Overall positive and negative emotions ratio can also be created by computing the mean of 10 positive emotions divided by mean of 10 negative emotions. The scale is suitable to be used with adolescents

SECONDARY OUTCOMES:
Daily Hassles | 4 weeks
  Daily Hassles: It is assessed through Inventory of High-School Students' Recent Life Experiences (IHSSRLE) is a self-reported reliable and valid measure that assesses daily hassles among adolescents.The scale has been developed by Kohn and Milrose in 1993. The inventory has 41 items with four points scoring ranging from 01(Not at all) to 04 (Completely true) and has eight (08) subscales. A high score reflects a high-stress level.

CONTACTS AND LOCATIONS:
Locations (1):
- Govt Islamia High School & Govt Girls High School, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
In SPSS sheet, Alpha Numerical ID will be assigned to each participant and only the combined statistical results would be published.